CLINICAL TRIAL: NCT01285661
Title: Identification of the Optimal Duration of Anticoagulation in Patients With Deep Venous Thrombosis of the Lower Extremities With the Use of Residual Vein Thrombosis in Combination With D-Dimer
Brief Title: Optimal Duration of Anticoagulation in Deep Venous Thrombosis
Acronym: MORGAGNI
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Padova (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2001P
Record Dates: First submitted 2010-04-30; First posted 2011-01-28 (Estimated); Last update posted 2016-07-19 (Estimated); Status verified 2016-07

CONDITIONS: Deep Vein Thrombosis of Lower Limb; Lower Extremity Deep Venous Thrombosis Recurrent
Keywords: Deep venous thrombosis; Pulmonary embolism; Ultrasonography; D-dimer; Venous thromboembolism; Bleeding
MeSH Terms: conditions — Venous Thrombosis; Pulmonary Embolism; Venous Thromboembolism; Hemorrhage | interventions — Vitamin B 6; acarboxyprothrombin; Anticoagulants

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Proximal DVT (Experimental): Patients whose veins have recanalized (either at the recruitment or later on during the follow-up) will receive the D-dimer determination before discontinuing sodium warfarin. Veins are defined as recanalized when the vein diameter under maximum compressibility is lower than 4 mm both at the common femoral and at the popliteal vein. In those with negative D-dimer sodium warfarin will be discontinued. These patients will have two further determinations of D-dimer (after 1 and 3 months, respectively). While patients with persistently negative D-dimer will no longer receive sodium warfarin, those in whom D-dimer is positive or reverts to positive values in the following determinations will have their sodium warfarin resumed and no longer discontinued.
  Interventions: Drug: Sodium warfarin

INTERVENTIONS:
Drug: Sodium warfarin — Patients with early vein recanalization, as shown by ultrasonography, and repeatedly negative D-dimer will have anticoagulation discontinued. They will be followed-up for up to 4 years after recruitment in order to assess the rate of recurrent symptomatic VTE. In all other patients anticoagulation will not be discontinued.
  Other Names: Vitamin K antagonists; Oral anticoagulants

SUMMARY:
Prospective cohort study aimed at optimizing the duration of anticoagulant treatment in patients at their first episode of proximal deep venous thrombosis (DVT) of the lower extremities, whose pathogenesis is either unknown (idiopathic DVT) or associated with minimal risk factors for thrombosis, with the help of an algorithm which incorporates both ultrasonography and D-dimer information. All patients will be followed-up until 1) the achievement of a major end-point; 2) the date of lost to to followup; 3) the date of death; 4) the date of study stop. The purpose of this study is to demonstrate the safety of withholding anticoagulation from a subgroup of patients with proximal DVT whose veins have recanalized and present with a repeatedly negative D-dimer (at baseline, after 1 and 3 months). The approach will be deemed to be safe if the annual rate of recurrent VTE in patients who will have their anticoagulation discontinued is lower than 5%.

DETAILED DESCRIPTION:
After giving informed consent, patients will receive an ultrasound investigation of the proximal-vein system (common femoral vein at groin, popliteal vein up to its trifurcation):

* Patients with residual thrombosis (defined as a diameter of at least 4 mm in at least one spot) will have their anticoagulation continued. A repeat ultrasound is scheduled after 6, 12, 18, 24 and 36 months. In patients with persistently residual thrombosis anticoagulation will not be discontinued, while those whose veins have recanalized will have a decision making process based on the behaviour of D-dimer (see below).
* Patients whose veins have recanalized (either at the recruitment or later on) will receive the D-dimer determination before discontinuing anticoagulation. In those with negative D-dimer anticoagulation will be discontinued. These patients will have two further determinations of D-dimer (after 1 and 3 months, respectively). While patients with persistently negative D-dimer will no longer receive anticoagulation, those in whom D-dimer becomes positive will have their anticoagulation resumed and no longer discontinued.
* All patients will be followed up to completion of 4 years since recruitment. For the purpose of this study each quantitative D-dimer is allowed. The criterion for D-dimer interpretation will rely on the cut-off that is recommended by manufacturers for diagnostic purposes.

D-dimer.For the purpose of this study each quantitative D-dimer is allowed. The criterion for D-dimer interpretation will rely on the cut-off that is recommended by manufacturers for diagnostic purposes.

Sample size 1000 years of observation without anticoagulation are required to demonstrate (power 90%, type I error 0.05, two sided) that with this approach the annual rate of recurrent VTE is lower than 5%. Approximately 600 patients with proximal DVT satisfying the eligibility criteria are required to obtain 1000 years of observation without anticoagulation.

ELIGIBILITY:
Inclusion Criteria:

* Patients with proximal DVT that is idiopathic or secondary to minor factors for thrombosis, with or without contemporary manifestations of PE, who have completed an uneventful 3 to 24-month period of anticoagulation and are available for an overall 48-month follow-up at the study centre.

Exclusion Criteria:

* previous thromboembolism
* recent (less than 3 months) major trauma or surgery
* active cancer
* immobilization resulting from chronic irreversible medical diseases
* need for indefinite anticoagulation for medical reasons other than VTE
* impossibility to attend the follow-up visits or to have D-dimer determinations
* already known major thrombophilia: carriage of deficiencies of natural anticoagulants, lupus-like anticoagulants, homozygosis for factor V Leiden or prothrombin mutation, heterozygosis for both abnormalities
* short (less than 1 year) life expectancy
* pregnancy
* age younger than 18
* refusal of informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 584 (Actual)
Dates: Start 2010-03; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Recurrent venous thromboembolism (VTE) | Up to the study conclusion (see the study protocol)
  To assess the rate of recurrent symptomatic VTE (expressed as rate/1000 patients-yeas) occurring after discontinuation of oral anticoagulant therapy up to the study conclusion.

SECONDARY OUTCOMES:
Development of major bleeding complications | Up to the study conclusion (see the study protocol)
  To assess the rate of major or clinically relevant bleeding complications (expressed as rate/1000 patients-years) occurring during oral anticoagilant therapy up to the study conclusion

CONTACTS AND LOCATIONS:
Overall Officials: Paolo Prandoni, Principal Investigator — Department of Cardiothoracic and Vascular Sciences, University of Padua
Locations (1):
- Paolo Prandoni, Padua, Italy

REFERENCES:
- [Derived] Prandoni P, Vedovetto V, Ciammaichella M, Bucherini E, Corradini S, Enea I, Cosmi B, Mumoli N, Visona A, Barillari G, Bova C, Quintavalla R, Zanatta N, Pedrini S, Villalta S, Camporese G, Testa S, Parisi R, Becattini C, Cuppini S, Pengo V, Palareti G; Morgagni Investigators. Residual vein thrombosis and serial D-dimer for the long-term management of patients with deep venous thrombosis. Thromb Res. 2017 Jun;154:35-41. doi: 10.1016/j.thromres.2017.04.002. Epub 2017 Apr 4. PMID 28407492